CLINICAL TRIAL: NCT03464760
Title: Evaluation of the Effect of Spirulina-Silicon Supplementation on the Morphological, Biomechanical and Functional Characteristics of the Arterial Wall in the Elderly
Acronym: ANGIO SPIRUL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Phyco-Biotech (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LOCAL/2016/APM-01; 2017-A00981-52 (Other: ANSM)
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2023-10

CONDITIONS: Elderly
MeSH Terms: interventions — Silicones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo
- Spirulina-Silicon supplementation (Experimental)
  Interventions: Dietary Supplement: 3.5g of spirulina per day in 1% silicone

INTERVENTIONS:
Dietary Supplement: 3.5g of spirulina per day in 1% silicone — 5 tablets of 700mg per day
  Arms: Spirulina-Silicon supplementation
Dietary Supplement: placebo — 5 tablets per day of potato-based placebo
  Arms: Placebo

SUMMARY:
The investigators hypothesize that spirulina-silicon supplementation will lead to an improvement in vasomotor endothelial function, followed by decreased arterial wave velocity on the aorta and central arterial pressure compared to placebo subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have given their free and informed consent and signed the consent form
* The subject must be a member or beneficiary of a health insurance plan
* The subject is available for 6 months of follow-up
* The subject must not have any pre-existing chronic illness nor any revealed during the pre-inclusion visit, either treated or requiring treatment according to current recommendations

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Presence of a chronic cardio-vascular and/or metabolic illness, known or revealed by the pre-inclusion exam and requiring treatment in accordance to official recommendations (HAS)
* Any other chronic pathology requiring medical treatment
* History of uric acid metabolism disorders (hyperuricemia, gout, urolithiasis).
* Subject presenting a loss of limitation of autonomy
* Treated with hormone replacement therapy in females
* Active smoker or drug user
* Presence of an abnormality revealed by the pre-inclusion biological assessment of dyslipidemia justifying a prescription medication, diabetes or intolerance to glucose (insulin resistance).
* Presence of a stenosis (greater than 50% in diameter, NASCET method) or carotid occlusion revealed by the echo-Doppler screening test.
* Presence of an aneurysm (dilation> 30 mm) of the abdominal aorta revealed by the echo-Doppler screening test.
* Arteriopathy of the lower limbs (toe systolic pressure (tsp) <0.7) revealed by the screening test (SysToe™ device).
* Subject already taking a food supplement based on spirulina or silicon.
* History of cardio-vascular disease or heart attack
* Subject develops a chronic illness requiring medical treatment for more than 7 days or a surgical intervention leading to incapacity for more than 7 days,or a pathological event during the 14-day period before each follow-up visit, or a serious adverse event

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Arterial Pressure Waveforms between groups | Month 6
  Applanation tonometry; m.s-1

SECONDARY OUTCOMES:
Arterial Pressure Waveforms between groups | Day 0
  Applanation tonometry; mm
Arterial Pressure Waveforms between groups | Month 1
  Applanation tonometry; mm
Arterial Pressure Waveforms between groups | Month 3
  Applanation tonometry; mm
Vasomotor endothelial function between groups | Day 0
  % post-ischemic vasorelaxation
Vasomotor endothelial function between groups | Month 1
  % post-ischemic vasorelaxation
Vasomotor endothelial function between groups | Month 3
  % post-ischemic vasorelaxation
Vasomotor endothelial function between groups | Month 6
  % post-ischemic vasorelaxation
intima-media thickness of common carotid arteries | Day 0
  echography; mm
intima-media thickness of common carotid arteries | Month 6
  echography; mm
left ventricular diastolic function | Day 0
  kPa
left ventricular diastolic function | Month 6
  kPa
Central venous pressure | Day 0
  mmHg
Central venous pressure | Month 1
  mmHg
Central venous pressure | Month 3
  mmHg
Central venous pressure | Month 6
  mmHg
Arterial Pressure Waveforms of females compared to males | Month 6
  Applanation tonometry; m.s-1
Vasomotor endothelial function of females compared to males | Month 6
  % post-ischemic vasorelaxation
Bone density | Day 0
  dual-photon absorptiometry
Bone density | Month 6
  dual-photon absorptiometry
Biological markers of vascular remodeling, oxidative stress and inflammation | Day 0
  Total cholesterol, High density lipoproteins, Triglycerides, Complete Blood Count, high-sensitivity C-reactive protein, toe systolic pressure, Oxidized low density lipoprotein, Vitamin E, Vitamin C, Reduced (GSH) and Oxidized (GSSG) Glutathione ratio, Procollagen type I N propeptide, cross-linking telopeptide of type I collagen, Elastin, Osteoprotegerin, Sclerotin, Calcium, Phosphorus, Alkaline Bone Phosphatase
Biological markers of vascular remodeling, oxidative stress and inflammation | Month 6
  Total cholesterol, High density lipoproteins, Triglycerides, Complete Blood Count, high-sensitivity C-reactive protein, IsoP, Oxidized low density lipoprotein, Vitamin E, Vitamin C, Reduced (GSH) and Oxidized (GSSG) Glutathione ratio, Procollagen type I N propeptide, cross-linking telopeptide of type I collagen, Elastin, Osteoprotegerin, Sclerotin, Calcium, Phosphorus, Alkaline Bone Phosphatase

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Perez-Martin, MD, Principal Investigator — CHU Nimes
Locations (1):
- CHU Nimes, Nîmes, France

REFERENCES:
- [Result] Virsolvy A, Benmira AM, Allal S, Demattei C, Sutra T, Cristol JP, Jouy N, Richard S, Perez-Martin A. Benefits of Dietary Supplementation with Specific Silicon-Enriched Spirulina on Arterial Function in Healthy Elderly Individuals: A Randomized, Placebo-Controlled Trial. Nutrients. 2025 Feb 28;17(5):864. doi: 10.3390/nu17050864. PMID 40077730